CLINICAL TRIAL: NCT06074965
Title: The Impact of Two Medtronic Infusion Sets (a 3-day Set & a 7-day Set) on Lipohyperthrophy (LH) in Persons With Type 1 Diabetes (T1D) and Thought to Have LH
Brief Title: Impact of Two Medtronic Infusion Sets on Lipohypertrophy in Type 1 Diabetes (T1DM) Patients Thought to Have LH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera San Camillo Forlanini (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Claudio Tubili, Head of Diabetology, Azienda Ospedaliera San Camillo Forlanini
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 299_CELazio1_220322
Record Dates: First submitted 2023-09-18; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Lipohypertrophy
Keywords: Lipohypertrophy; Infusion Sets; Insulin Pump; CGM
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This is a 1-center, prospective, open label, 2-arm study of ≥16 subjects who use the insulin pumps. These subjects will be using 2 types of infusion sets for two periods of 3 months each type that will serve as an exploratory pilot study to assess the impact of infusion sets on lipohypertrophy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): These subjects will be using infusion set A for the first 3 months and infusion set B for the following 3 months
  Interventions: Device: Medtronic Extended Infusion Set
- Arm 2 (Experimental): These subjects will be using infusion set B for the first 3 months and infusion set A for the following 3 months
  Interventions: Device: Medtronic Extended Infusion Set

INTERVENTIONS:
Device: Medtronic Extended Infusion Set — Each subject will be given 2 types of infusion sets to wear and change sets per label use (3 days for Medtronic Quick-set™ and 7 days for Medtronic Extended).
  Other Names: Medtronic Quick-set™ Infusion Set

SUMMARY:
This is an observational study using ultrasound (US) and palpation to assess the impact of infusion sets on lipohypertrophy (LH) in an infusion set crossover study.

DETAILED DESCRIPTION:
This is a 1-center, prospective, open label, 2-arm study of ≥16 subjects who use the insulin pumps. These subjects will be using 2 types of infusion sets for two periods of 3 months each type that will serve as an exploratory pilot study to assess the impact of infusion sets on Lipohypertrophy LH (see Figure 1 for study design).

Each subject will use their own MiniMed™ 670G insulin system as usual. Each subject will be given 2 types of infusion sets to wear and change sets per label use (3 days for Quick-set™ and 7 days for Medtronic Extended). Each type of infusion set with the longest length (43" in) will be used for this study. 7-day reservoirs will be used with the Medtronic Extended and 3-day reservoirs will be used with the Quick-set™. The infusion set(s) or reservoir(s) can be replaced independent of each other for Medtronic Extended.

The subject will use either Medtronic Extended or Quick-set™ infusion set for consecutive 3 months. During the three-month period, either the right side or the left side of the abdomen will be designated for one or the other infusion set (defined randomly). For each type of infusion set, a coordinate rule for site rotation will be given to have the Set placed in a specified area (left or right side) of anterior abdominal wall.

For each placement/wear, a daily log will be given to the subject to record time and location for the infusion set placement. Patients will be instructed to recognize areas of clinical apparent LH sites and refrain from inserting in these areas. At home, the subject will be expected to inspect their infusion site on a daily basis and if they observe signs of infection (i.e. erythema > 1 cm in diameter with warmth, pain, and/ or induration) at the infusion site, they should call the investigational center. In addition to the study procedures, the subjects are to continue their standard routine care. In the end of each month, the subject should self-inspected by palpation for LH and record the findings on the daily log.

At each study visit, insulin pump and CONTOUR® NEXT LINK 2.4 study meter will be uploaded into CareLink™ Personal For Clinical Research. Also, all the infusion sites will be examined ultrasonically for LH.

At each visit the clinical team will assess the skin in a systematic using the palpation method procedure and the ultrasound (US) evaluation procedure.

All participants will be asked to give demographic details and medical history. They will be asked to complete a series of questionnaires about their pump routine, diabetes distress, insulin treatment satisfaction and quality of life. All participants will have a baseline glycated hemoglobin (HbA1C) taken. The Total Daily Dose (TDD) will be calculated based on the CareLink™ data.

It is anticipated that approximately 16 subjects will complete the study and up to 20 subjects may be screened. As this is an exploratory study, no power assumptions are planned. The study is anticipated to last up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes and has been a pump user for at least 10 years
* Using a MiniMed™ 670G or 640G Insulin pump with Guardian sensor
* Age 18 to 80 years
* Hemoglobin A1c level less than or equal to 10%
* Not currently known to be pregnant, nor planning pregnancy during the study.
* Willingness to follow the protocol and sign the informed consent
* Use U100 Humalog (insulin lispro) or U100 NovoRapid/Novolog (insulin aspart)

Exclusion Criteria:

* Conditions that affect the skin evaluation, e.g. scleroderma or amyloidosis
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.
* Pregnant or lactating females
* Subject has Glycosylated hemoglobin (HbA1c) > 10 % at time of screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Event rate of lipohypertrophy (LH) | 6 months
  The study will be evaluated and summarized, including but not limited to the following:
  * Self-assessed LH by palpation using a visual analogue scale (VAS) 1 to 10, coupled with clinical examination by a physician if possible.
  * LH (appearance, location, mass, indices of vascularization and distribution) characterized by ultrasound.
  * The relationship between the observed LH and infusion set type, TDD, glycemic control, HbA1C etc.
  * Satisfaction of infusion sets using validated questionnaire, e.g. the diabetes treatment satisfaction questionnaire (DTSQ).

SECONDARY OUTCOMES:
Continuous Glucose Monitoring (CGM) data: Time Above Range (TAR) | 6 months
  Duration, and area under the curve (AUC) when Sensor Glucose>180, >240, and >250 mg/dL
Continuous Glucose Monitoring (CGM) data: Time Below Range (TBR) | 6 months
  Duration, area under the curve (AUC) when Sensor Glucose <50, <60, and <70 mg/
Continuous Glucose Monitoring (CGM) data: Time In Range (TIR) | 6 months
  Duration, area under the curve (AUC) when Sensor Glucose > 70 e < 180 mg/dL
Glycemic variability: Standard Deviation (SD), Coefficient of Variation (CV), mean amplitude of glycemic excursions (MAGE) | 6 months
Cohort analysis by age | 6 months
Cohort analysis by duration of diabetes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Tubili, Principal Investigator — Azienda Ospedaliera San Camillo Forlanini
Locations (1):
- Azienda Ospedaliera San Camillo Forlanini, Roma, Italy

DOCUMENTS (1):
  • Study Protocol (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT06074965/Prot_000.pdf